CLINICAL TRIAL: NCT02906098
Title: A Randomized Clinical Field Study on Behavioral Interventions to Increase Adolescent's Motivation for Self Performed Periodontal Infection Control
Brief Title: Intervention Study of Oral Health Education Programs Directed to Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: kajsaha
Record Dates: First submitted 2016-09-07; First posted 2016-09-19 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Gingivitis; Periodontal Infection
Keywords: Gingivitis; Adolescents; Oral hygiene; Oral health behavior; Periodontal infection control
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient centered oral health education (Experimental): The program is based on cognitive behavioral theory and principles. Hence, the intervention is adapted to each individual's problem, capacity and goals were the dental hygienist use motivational interviewing skills in communication and act as a guiding resource during the process of behavioral change. The program follows a specific structure including components such as formulation of personal goals, continuous self-monitoring by diary and planning of behavior. The initial intervention phase contain 3 treatment sessions (45-60 min each) during a period of 12 weeks (baseline, 2-3 weeks and 10-12 weeks). Follow up are performed at 6- and 18-months.
  Interventions: Behavioral: Patient centered oral health education
- Standard educational intervention (Active Comparator): The subjects in the control group receive educational intervention by a dental hygienist in accordance with conventional routines (oral health information and oral hygiene instruction at one or several occasions). Follow up are performed at 6- and 18-months.
  Interventions: Behavioral: Standard educational intervention

INTERVENTIONS:
Behavioral: Patient centered oral health education — Procedure: The theory-based educational intervention follows a specific structure. The initial phase contain 3 treatment sessions (45-60 min each) during a period of 12 weeks (baseline, 2-3 weeks and 10-12 weeks). Follow up are performed at 6- and 18-months.
  Arms: Patient centered oral health education
Behavioral: Standard educational intervention — Procedure: The initial phase contain educational intervention in accordance with conventional routines (oral health information and oral hygiene instruction at one or several occasions). Follow up are performed at 6- and 18-months.
  Arms: Standard educational intervention

SUMMARY:
This study evaluates behavioral interventions to increase adolescent's motivation for self performed periodontal infection control, by means of adequate oral hygiene. Study subjects will be allocated to test and control group where the test will be subjected to an individually tailored oral health education program, based on cognitive- behavioral theory and principles, and the control to standard educational intervention.

DETAILED DESCRIPTION:
The prevalence of chronic periodontitis is about 40% among the Swedish adult population. The key-factor for the prevention of periodontal disease progression is the establishment of periodontal infection control, by means of adequate daily oral hygiene. Hence, a main task for dental professionals is to educate and motivate the patient to such beneficial behavior. A hypothesis for the current study is that patient centered health promotion programs based on cognitive behavioral theory and principles and with a directive communicative approach, i.e. motivational interviewing techniques, add positive and lasting effects to standard educational interventions on self-performed periodontal infection control.

This randomized clinical field study involves 30 professionals (dental hygienists) and about 350 adolescent patients at 16 dental clinics in the Västra Götaland Region, Sweden. The approach in the evaluation is on patient-centered outcomes and health economics.

ELIGIBILITY:
Inclusion Criteria:

* 16 or 17 years old at inclusion
* poor oral hygiene conditions (dental plaque and/or marginal gingival bleeding at >50% of tooth surfaces) at the time of examination and thus considered to be at increased risk for oral/periodontal disease progression.

Exclusion Criteria:

* compromised medical or mental conditions that may requiring special care.

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 312 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Marginal gingival bleeding index | Up to 18-months
  Percentage of tooth-surfaces with bleeding (infection) at clinical examination

SECONDARY OUTCOMES:
Patient reported outcome measures (PROM) | Up to 18-months
  Questionnaire
Patient reported experience measures (PREM) | Up to 18-months
  Questionnaire
Individual investment for treatment - Direct and subsidiary costs | Up to 18-months
  Questionnaire - time, travel costs, costs for potential accompanying person

OTHER OUTCOMES:
Plaque score | Up to 18-months
  Percentage of tooth-surfaces with dental plaque at clinical examination
Treatment time for behavioral intervention in relation to total treatment time | Up to 18-months
  Questionnaire - assessment by caregiver regarding different treatment procedures

CONTACTS AND LOCATIONS:
Overall Officials: Kajsa H Abrahamsson, Odont Dr, Principal Investigator — Dept of periodontology, Inst of odontology, The Sahlgrenska academy, University of Gothenburg
Locations (1):
- Kajsa H Abrahamsson, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dimenas SL, Ostberg AL, Lundin M, Lundgren J, Abrahamsson KH. Adolescents' experiences of a theory-based behavioural intervention for improved oral hygiene: A qualitative interview study. Int J Dent Hyg. 2022 Nov;20(4):609-619. doi: 10.1111/idh.12606. Epub 2022 Aug 15. PMID 35925040
- [Derived] Dimenas SL, Jonsson B, Andersson JS, Lundgren J, Petzold M, Abrahamsson I, Abrahamsson KH. A person-centred, theory-based, behavioural intervention programme for improved oral hygiene in adolescents: A randomized clinical field study. J Clin Periodontol. 2022 Apr;49(4):378-387. doi: 10.1111/jcpe.13601. Epub 2022 Feb 23. PMID 35132653